CLINICAL TRIAL: NCT00205023
Title: The Incidence of Disseminated Endometrial Cancer Cells During Sonohysterography and Their Functional Viability: a Prospective Study
Brief Title: Disseminated Endometrial Cancer Cells During Sonohysterography
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CO03702; H-2003-0499 (Other: Institutional Review Board); A532820 (Other: UW Madison); SMPH/OBSTET & GYNECOL (Other: UW Madison)
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2019-11-19 (Actual); Status verified 2008-06

CONDITIONS: Endometrial Cancer
MeSH Terms: conditions — Endometrial Neoplasms

ARMS (1):
- A (Experimental)
  Interventions: Procedure: Sonohysterography

INTERVENTIONS:
Procedure: Sonohysterography — SHG during surgery for endometrial cancer.

SUMMARY:
The purpose of study is to: 1) determine critical volume necessary to overcome tubal pressure and result in fluid dissemination and 2) evaluate functional viability of any disseminated tumor cells collected during SHG

ELIGIBILITY:
Inclusion Criteria:

* Stage I endometrial Cancer Disease
* State IIA endometrial Cancer Disease

Exclusion Criteria:

* Prior tubal ligation
* Prior bilateral salpingectomy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2004-01; Primary Completion 2006-02 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
determine the critical volume necessary to overcome tubal pressure and result in fluid dissemination during SHG | during surgery

SECONDARY OUTCOMES:
evaluate the functional viability of any disseminated tumor cells collected during SHG | during surgery

CONTACTS AND LOCATIONS:
Overall Officials: David M Kushner, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

REFERENCES:
- See also: University of Wisconsin Carbone Cancer Center — https://cancer.wisc.edu